CLINICAL TRIAL: NCT05996679
Title: Automated Surveillance, Alert, and Rapid Diagnosis of Thrombotic Microangiopathies: the ASARD-TMA Study
Acronym: ASARD-TMA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, DE STEFANO VALERIO, Full Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 5761
Record Dates: First submitted 2023-08-10; First posted 2023-08-18 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Thrombotic Microangiopathies
MeSH Terms: conditions — Thrombotic Microangiopathies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Recently a pilot study was conducted to evaluate the impact of an electronic alert (e-alert) triggered by the automated algorithm in the efficiency and rapidity in TMA patients' identification in our University Hospital A. Gemelli over 12 months.the TMA diagnostic algorithm has been implemented in the laboratory software of the hospital and applied whenever a patient in the Emergency ward or any other department undergoes blood tests that include platelet count and lactate dehydrogenase. The basic profile in the Emergency ward always has these two parameters. The algorithm automatically identifies patients with a predicted probability of TMA >90% (6); if this criterion is associated with a platelet count<100 x 109/L, an automated warning to the hematologist on-call is issued with an SMS, and the patient enters the TMA diagnostic process defined in the diagnostic and treatment pathways (Percorso Diagnostico e Terapeutico Assistensiale, PDTA). The on-duty hematologist urgently evaluates the patient for whom a warning has been issued, relating with the clinician(s) of the ward in which the patient is located. If the suspicion of TMA is confirmed, the diagnostic procedures outlined in the PDTA are performed, with the immediate execution of 2nd level tests. If the on-duty hematologist considers the diagnosis of aHUS possible, they contact the on-call Nephrologist directly for immediate diagnostic investigation and specific urgent therapeutic measures, as needed. The TMA-expert Hematologist and/or TMA-expert Nephrologist is notified as soon as possible by the on-duty hematologist of all cases, both highly suspected and uncertain, and follow up all patients to complete the diagnostic workup to confirm or rule out the diagnosis and implement the appropriate clinical measures.

Therefore, the treatment in smaller hospitals that do not have a 24-hour hematological guard service available and the same awareness for TMA.

The present study aims to validate these results by testing the system in a multicenter study involving centers with different availability of the hematologist and awareness for TMA.

ELIGIBILITY:
Inclusion Criteria:

Patients admitted to the Emergency ward or inpatients of the involved Hospitals with suspicion of TMA:

* Based on the clinical evaluation of the care physicians
* Based on the alerts issued by the automated algorithm

Exclusion Criteria:

* Patients with a predictive probability of TMA < 90% (6) according to the diagnostic algorithm

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study will be conducted in 4 Hospitals (Nefrologia e Dialisi Ospedale Maggiore Verona; Area Aggregata di Ematologia, Fondazione Policlinico Tor Vergata, Roma; Nefrologia e Dialisi ASST Santi Paolo e Carlo, Università di Milano; Nefrologia e Dialisi AOU G. Martino - Università degli Studi di Messina) over 12 months.
Sampling Method: Probability Sample
Enrollment: 29 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Time of diagnosis and treatment of Thrombotic microangiopathies | 24 months
  Evaluating algorithm to speed up diagnosis and treatment of TMA in smaller hospitals that do not have a 24-hour hematological guard service available and the same awareness for TMA.